CLINICAL TRIAL: NCT04932213
Title: Comparison of the Effect of Tropicamide 0.5% and Tropicamide 1% on Intraocular Pressure, Pupil Size, Keratometry and Anterior Chamber Parameters in Patients With Type 1 and Type 2 Diabetes Mellitus
Brief Title: Effect of Tropicamide 0.5% vs Tropicamide 1% on Intraocular Pressure of Diabetic Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Semnan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Navid Elmi Sadr, Assistant professor of ophthalmology, Semnan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IR.SEMUMS.REC.1400.018; IRCT (Registry Identifier: IRCT20200829048553N1)
Record Dates: First submitted 2021-06-07; First posted 2021-06-21 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Type 2 Diabetes Mellitus; Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Intervention group 1: This group receives tropicamide 0.5% drops; Intervention group 2: This group receives tropicamide 1% drops.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The drops are instilled into the patients' eye by a nurse. Study participants are unaware of the type of medication used. The outcome assessor (ophthalmologist) does not know the type of medication used for each patient. The data is analyzed by an biostatistician. He or she also does not know the type of drug used for each patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tropicamide 0.5% (Active Comparator): This group receives tropicamide 0.5% (one drop every 5 minutes for 2 times) drops.
  Interventions: Drug: Tropicamide Ophthalmic
- Tropicamide 1% (Active Comparator): This group receives tropicamide 1% (one drop every 5 minutes for 2 times) drops.
  Interventions: Drug: Tropicamide Ophthalmic

INTERVENTIONS:
Drug: Tropicamide Ophthalmic — Tropicamide eye drops are used for dilating pupils (mydriasis) to do comprehensive fundus examination.
  Other Names: Mydrax (Sina Darou)

SUMMARY:
The aim of this study is to compare the effect of tropicamide 0.5% and tropicamide 1% on intraocular pressure and anterior chamber parameters in patients with Diabetes Mellitus.

DETAILED DESCRIPTION:
Patients with diabetes type 1 and type 2 older than 21 years of age, in the specialized clinic of Kowsar Hospital (Semnan University of Medical Sciences) are examined. Eligible individuals enter the study and are randomly assigned to group 1 or group 2. In each group, visual acuity measurement, slit lamp biomicroscopy and fundus examination are performed. Intraocular pressure is measured with Goldmann applanation tonometer. pupil size, refraction and keratometry are measured with two different autorefractokeratometers. keratometry, pupil size and other anterior chamber parameters are also evaluated by Oculus Pentacam imaging. Then, the patients receive tropicamide 0.5% drops in group 1 and tropicamide 1% drops in group 2. 30 minutes later, all previous measurements are repeated. Patients and the ophthalmologist and the data analyzer are unaware of the drug type.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Diabetes Mellitus type 1 and 2

Exclusion Criteria:

* Proliferative diabetic retinopathy
* History of cataract surgery
* severe nuclear and cortical cataract
* Glaucoma
* Intraocular pressure (IOP) greater than 21 mmHg
* Familial history of glaucoma
* Narrow angle (Van Herick 1, 2)
* Cup to disc ratio greater than 0.5
* Pregnancy
* Pterygium
* Corneal ectasia
* History of keratorefractive surgery
* Corneal dystrophy
* Iris disorders
* Anisocoria
* Iris neovascularization
* Use of miotics or mydriatics

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-11-07 (Actual); Study Completion 2021-11-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Intraocular pressure (IOP) | Before intervention, 30 minutes after intervention
  The intraocular pressure is measured by Goldmann applanation tonometry
Change from baseline in pupillary diameter | Before intervention, 30 minutes after intervention
  The diameter of the participants' pupil is measured by Scheimpflug camera (Oculus Pentacam); Autorefractokeratometer (TOMEY RC-5000 and Topcon KR-1)

SECONDARY OUTCOMES:
Change from baseline in Keratometry | Before intervention, 30 minutes after intervention
  The keratometry is obtained by Scheimpflug camera (Oculus Pentacam); Autorefractokeratometer (TOMEY RC-5000 and Topcon KR-1)
Change from baseline in anterior chamber depth (ACD) | Before intervention, 30 minutes after intervention
  The ACD is measured by Scheimpflug camera (Oculus Pentacam)
Change from baseline in anterior chamber volume (ACV) | Before intervention, 30 minutes after intervention
  The ACV is measured by Scheimpflug camera (Oculus Pentacam)
Change from baseline in anterior chamber angle (ACA) | Before intervention, 30 minutes after intervention
  The ACA is measured by Scheimpflug camera (Oculus Pentacam)
Change from baseline in central corneal thickness (CCT) | Before intervention, 30 minutes after intervention
  The CCT is measured by Scheimpflug camera (Oculus Pentacam)

CONTACTS AND LOCATIONS:
Overall Officials: Navid Elmi Sadr, MD, Principal Investigator — Semnan University of Medical Sciences, Semnan, Iran; Navid Elmi Sadr, MD, Study Director — Semnan University of Medical Sciences, Semnan, Iran
Locations (1):
- Kowsar Semnan Research and Medical Training Center, Semnan, Iran

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared without disclosing the identities of the participants.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Access period starts one year after the results are published.
Access Criteria: Researchers can use the data for systematic review studies and meta-analysis. Researchers working in academic and scientific institutions can contact the person in charge of the scientific inquiries of the project by e-mail. After receiving the request e-mail, if the person is eligible, the data will be sent